CLINICAL TRIAL: NCT03253640
Title: Evaluation of Cost of Nosocomial Infection
Acronym: ECONI
Status: Completed | Type: Observational
Sponsor: Glasgow Caledonian University (Other)
Collaborators: University of Strathclyde (Other); Nick Graves Independent Consultant (Unknown); NHS Lothian (Other Government); NHS Lanarkshire (Other Government)
Responsible Party: Sponsor
Other Study IDs: 14-154; IRAS Identifier (Other: Integrated Research Application System)
Record Dates: First submitted 2017-02-24; First posted 2017-08-18 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-01

CONDITIONS: Crossing Infections; Drug Resistance, Microbial
Keywords: Costs and Cost Analysis; Quality of Life; Length of Stay; Cohort study
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with HAI during hospital stay: Patients who meet the European Centre for Disease Control (ECDC) Healthcare Associated Infection (HAI) case definitions. Case note review will be undertaken during hospital stay. Questionnaire will be administered at recruitment, pre-discharge, one, three, six and twelve months post discharge.
  Interventions: Other: Exposure
- Patients without HAI during hospital stay: Patients who do not meet the European Centre for Disease Control (ECDC) Healthcare Associated Infection (HAI) case definitions. Case note review will be undertaken during hospital stay. Questionnaire will be administered at recruitment, pre-discharge, one, three, six and twelve months post discharge.

INTERVENTIONS:
Other: Exposure — Healthcare associated infection (HAI)
  Groups: Patients with HAI during hospital stay

SUMMARY:
This study will investigate the cost and impact of Healthcare Associated Infection (HAI) to patients, the health service and the wider community.

This is in order to develop a model to allow policy makers to compare the cost effectiveness of Infection Prevention and Control measures in NHSScotland. The model will support policy makers and clinical teams in building a patient centred, safe, effective and efficient service.

DETAILED DESCRIPTION:
Healthcare associated infection (HAI) also known as Nosocomial Infection (NI) is costly to the NHS and distressing to patients. It leads to increased morbidity and mortality, increased length of stay and often requires additional treatments. Information on the impact in terms of additional cost of treatment, reduction in quality of life and cost to society is not fully described. This study will collect epidemiological and economic data on patients with and without HAI and develop a framework around which the cost effectiveness of a range of Infection Prevention and Control (IPC) interventions can be assessed.

The study will be delivered as 4 distinct but overlapping work Phases Phase 1 will describe the incidence of HAI (defined by ECDC case definitions) in an admission cohort. This phase is a surveillance project.

Phase 2: Will describe the impact of HAI on care in hospital -as many patients as possible who acquired HAI and twice as many non-HAI comparators will be recruited. Patients or their guardians or nearest relative will be told about the study and asked if they are willing to provide consent to complete a number of questionnaires. This phase will include case note review by ECONI research nurses and a patient questionnaire.

Phase 3: Will investigate the impact of HAI on patient care post discharge (use of Health and Social Care resources outside of Hospital), Quality of Life and personal expenses) - questionnaire to patients to ask about impact on their overall health and wellbeing and personal expenses. This will involve patients completing a paper questionnaire at one, three, six and twelve months after they have been discharged from hospital. This phase will include a nested qualitative study which will interview 20-30 patients who acquired HAI to further investigate the impact of HAI on their lives and livelihoods Phase 4: This phase will not involve any patient interaction. It will develop a framework to support modelling for decision making for future investment in Infection Prevention and Control (IPC) based on data collected within Phase one to three above. The information collected during the first three phases will be used to model possible outcomes of infection prevention and control measures. This will be a modelling exercise using data collected within Phase 1, 2 and 3 and the protocol for this work will be described elsewhere.

Phase 2 and 3 will be a cohort of as many patients as possible with HAI and a sample of non-HAI patients (twice the number of HAI patients) who consent to participate in the study within the year of recruitment.

Modes of data collection

1. Research Nurse administered questionnaire on recruitment quality of life questionnaire on recruitment
2. Day before discharge quality of life questionnaire
3. 1 month post discharge questionnaire
4. 3 month post discharge questionnaire
5. 6 month post discharge questionnaire
6. 12 month post discharge questionnaire
7. Record linkage - SMOR00, SMR01, PRISMA, District nursing
8. 1,500-3,000 patients recruited for follow up.
9. All admissions to study hospitals for record linkage. Follow up duration 1 year post discharge from admission when patient was recruited.

Data will be collected using a Redcap database. Where possible controlled lists will be included within the database to ensure consistency of reporting. Validation visits to study sites will be undertaken throughout the study data collection period. Standard operating procedures will be developed for the ECONI team to use during recruitment and data collection. A data dictionary will be developed to record all data items recorded during the study, where these data were sourced, the choices available and the field-names within the data set. A publications and communication plan has been developed for the study and an analysis plan will be developed linking each of the objectives to a peer reviewed publication. A number of systematic reviews have be undertaken in the development of the ECONI study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to hospital for an overnight stay at study hospital
2. Subjects capable of giving informed consent, or if appropriate, subjects having an acceptable individual capable of giving consent on the subject's behalf
3. Any sex
4. 18 years old and over
5. Patients without HAI will not be re-recruited into the study. Patients who have HAI on a subsequent admission will not be re-recruited but will be asked to complete a baseline data collection form (see below for discussion) NOTE: we do need to ensure this is clear within the ethics application.
6. Good English language skills (sufficient to read and understand the participant information sheet without help)

Exclusion Criteria:

1. Admitted to hospital as a day case
2. Admitted to Hospitals other than the study hospitals
3. Under 18 years
4. Admitted to the study hospital during the study period and recruited to the study during a previous stay. See below
5. Subjects not capable of giving informed consent unless legal representative or relative can provide proxy consent
6. Patients who do not have English language skills to read and understand the information sheet without help

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to study hospitals over night during a one year study period
Sampling Method: Non-Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Acquisition of healthcare associated infection | During hospital stay, within one year post discharge for two hospital sites
  Number of patients who develop new HAI Defined using ECDC HAI case definitions, and including costs of care in hospital, post discharge and impact of usual activity, ability to work and social care.
Length of stay in hospital | All patient stays during the study year
  Date of admission to discharge
Healthcare utilisation | One year post discharge from hospital visit when recruited
  Includes, specialty, antibiotic use, operations, post discharge health visits, community prescribing, out patient clinic attendance, re-admission to hospital
Quality of Life | Utility score during hospital stay for HAI and non_HAI patients during hospital stay, one month post discharge and three months post discharge
  Quality of life will be measured using SF-12 and EQ-5D validated questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Jacqui M Reilly, PhD, Study Director — Glasgow Caledonian University
Locations (2):
- United Kingdom (2):
  - Hairmyres Hospital, East Kilbride
  - Edinburgh Royal Infirmary, Edinburgh

IPD SHARING:
Plan to Share IPD: Undecided
The study Steering Committee will review this at the end of the study. Data will be only be shared at an individual level if all identifiable information has been removed or categorised, individual records would be identified using a cypher code.

REFERENCES:
- [Derived] Stewart S, Robertson C, Manoukian S, Haahr L, Mason H, McFarland A, Dancer S, Cook B, Reilly J, Graves N; ECONI Steering Committee. How do we evaluate the cost of nosocomial infection? The ECONI protocol: an incidence study with nested case-control evaluating cost and quality of life. BMJ Open. 2019 Jun 19;9(6):e026687. doi: 10.1136/bmjopen-2018-026687. PMID 31221878